CLINICAL TRIAL: NCT03308500
Title: Effect of High-intensity Intermittent Games on Cardiorespiratory Fitness and Body Composition in Children
Acronym: HIIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Lusófona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LUSUP21231016
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Children, Physical Activity
Keywords: HIIT; Children; Cardiorespiratory fitness; Body composition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Experimental design is applied where HIIG is compared with MIG. The participants of the study will be divided into two groups; HIIG and MIG. Both of them will have two sessions per week during 12 weeks of intervention.
  Follow up: children are contacted 3 months after finishing the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity intermittent games HIIG (Experimental): High-intensity intermittent games (HIIG): complete a supervised 12-weeks. Twice per week child-specific games program, intensity HRmax 75% ≤ - RPE 6-8.
  Interventions: Behavioral: High-intensity intermittent games
- Moderate-intensity games (MIG) (Active Comparator): Moderate intensity games (MIG): complete a supervised 12-weeks. Twice per week child-specific games program, intensity HRmax 60-74% ≤ - RPE 4-5.
  Interventions: Behavioral: Moderate intensity games

INTERVENTIONS:
Behavioral: High-intensity intermittent games — The intervention will last for 12-weeks, each group included participation in twice-week 40 minutes exercise sessions. In HIIG children took part in 5 games per session; 2 velocity games and 3 small-sided games (such 3 vs 3 and 4 vs 4). This session included 4 minutes games and 2 minutes recovery. In MIG children took part in 5 games per session. This session included 4 minutes games and 3 minutes recovery.
  Arms: High-intensity intermittent games HIIG
Behavioral: Moderate intensity games — The intervention will last for 12-weeks, each group included participation in twice-week 40 minutes exercise sessions. In MIG children took part in 5 games per session. This session included 4 minutes games and 3 minutes recovery.
  Arms: Moderate-intensity games (MIG)

SUMMARY:
This study will assess the effectiveness of a high-intensity intermittent games intervention (HIIG) on cardiorespiratory fitness and corporal composition. Fifty-four children, aged 9-12 years, will be randomised into an HIIG or moderate-intensity games (MIG) group. Before and after the intervention, participants complete cardiorespiratory fitness and corporal composition test. The hypothesis states that there is an improvement in the cardiorespiratory fitness and in the body composition implementing high-intensity intermittent games.

DETAILED DESCRIPTION:
Background

Physical activity is associated with many health benefits, but most children fail to meet the international recommendation. This is a concerning matter for the future health-care population, as cardio-metabolic risk factors in children and adolescents can lead to coronary heart disease, metabolic diseases (obesity, type II diabetes) and mortality in adulthood.

According to children participated in different types of physical activity or early sports practice in the first stages of life has been positively associated with lower occurrence of chronic diseases in adulthood. Ultimately, daily participation in outdoor games, fitness activities, and recreational sports will be a major factor in the improvement of health and well-being of children and adolescents.

Unlike adults, children's habitual physical activity patterns are highly intermittent in nature, characterised by rapid changes from rest to vigorous physical activity.

High-intensity intermittent training (HIIT) describes physical exercise as a brief, intermittent burst of vigorous activity, interspersed by rest periods or low-intensity exercise. HIIT offers infinite variations with the specific physiological adaptations induced by this form of training determined by several factors including the precise nature of the exercise stimulus. In recent years HIIT has received great scientific interest, the studies have examined the physiological effects of HIIT in children and adolescents and reported positive findings on cardiorespiratory fitness, fat-free mass index, a change in body mass index (BMI) and percentage body fat.

Objective The objective of the study is to verify the effects of a high-intensity intermittent games intervention (HIIG) versus a moderate intensity group on cardiorespiratory fitness and body composition in children. The hypotheses formulated was: high-intensity intermittent games intervention contribute to the improvement cardiorespiratory fitness and body composition in children.

Methods

Study Setting This study is performed in a public school setting in the city of Valparaiso, Chile.

Participants timeline Will be recruited through information to the parents 54 children from 8 to 12 years old belonging to a public school of Valparaiso, Chile.

Interventions The intervention will last for 12-weeks, each group included participation in twice-week 40 minutes exercise sessions. In HIIG children took part in 5 games per session; 2 velocity games and 3 small-sided games (such 3 vs 3 and 4 vs 4). This session included 4 minutes games and 2 minutes recovery. In MIG children took part in 5 games per session. This session included 4 minutes games and 3 minutes recovery. A standardised warm-up protocol consisting of 5 minutes of running and stretching is performed before each training session. Cool down is after class 5 minutes of static stretching.

The intensity will be continuously monitored during each session through heart rate (Polar M400, Finland) and rating of perceived exertion (RPE). The intervention will be based on the protocols described by different authors of the area.

These sessions will be conducted inside of the children's normal physical education lessons. A Physical Education Professor will make the interventions. Thus, the study will be divided into four moments: T1 (recruitment and screening), T2 assessment before the intervention, and T3 and T4 for assessment after intervention and assessment follow up.

Sample size The sample is calculated a with variance analysis (ANOVA one way) (one independent variable) with an anticipated statistical power of 0.95, an error probability of 0.05, and effect size of 0.5, predicted that the appropriate sample size for the present study is 54 participants (G-power program 3.1.3, Germany).

The subject sample is comprised of 54 elementary school students aged 9-12 years. Participants and their parents had to sign a written consent containing all the information of the study prior to the commencing day.

Statistical analysis The normality distribution of the data will be checked with the Kolmogorov-Smirnov test. All data will be expressed as averages and standard deviations (DS).

ANOVA will be used to ensure that all 2 groups are homogeneous according to cardiorespiratory fitness and body composition before training.

The effects of training will be statistically analysed using post-hoc Tukey test in order to compare the variables present among the mean value groups between pre and post test (time effect). For each variable, there is an effect that could be attributed to the intervention or the gender. Therefore, in both groups, data for boys and girls will be collected and analysed by a 2-way ANOVA. The threshold for statistical significance is set at p ≤ 0.05. All analyses will be performed using Statistical Package for the Social Sciences (IBM SPSS) version 22.0.

The study contributes to scientific knowledge since it studies the effects of a new method of physical exercise which still lacks full clarity regarding its implementation and effect in variables like cardiorespiratory fitness and body composition in children.

The study is guided by practice-based scientific evidence for the use of HIIT in children. Upon completion of data collection, it is expected that the HIIG volunteers will benefit from increased cardiorespiratory fitness through the 20 meters shuttle run test, improved body composition through the decreased body fat mass and increased body muscle mass, reductions in scores on the IMC, and waist circumference. In the MIG, no significant changes in the values of any variable analysed are expected. It is believed that the desired results could be attributed to physiological effects of exercises of high-intensity intermittent exercises associated with the proposed exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

Children

Ages of 8 to 12

Tanner 1-2

Are not part of any regular exercise training program

Agree to the commitment

Exclusion Criteria:

Chronic paediatric disease (except for obesity)

Cardiovascular or metabolic disease

Orthopaedic limitation

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness; 20 meters shuttle run test | Pre - post intervention and follow up. Time which each participant is assessed; 40 minutes
  Maximum oxygen uptake (VO2max) metric: ml·kg-1·min-1

CONTACTS AND LOCATIONS:
Overall Officials: Tomás R Reyes, MSc, Principal Investigator — Faculty of Physical Education and Sport, University Lusofona/Faculty of Sciences Physical Activity and Sports, University Playa Ancha; Antonio L Palmeira, PhD, Study Director — Faculty of Physical Education and Sport, University Lusofona
Locations (1):
- University Playa Ancha, Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No
2 congresses 2 publications

REFERENCES:
- [Background] Lambrick D, Westrupp N, Kaufmann S, Stoner L, Faulkner J. The effectiveness of a high-intensity games intervention on improving indices of health in young children. J Sports Sci. 2016;34(3):190-8. doi: 10.1080/02640414.2015.1048521. Epub 2015 May 26. PMID 26009003
- [Background] Lee YH, Song YW, Kim HS, Lee SY, Jeong HS, Suh SH, Park JK, Jung JW, Kim NS, Noh CI, Hong YM. The effects of an exercise program on anthropometric, metabolic, and cardiovascular parameters in obese children. Korean Circ J. 2010 Apr;40(4):179-84. doi: 10.4070/kcj.2010.40.4.179. Epub 2010 Apr 23. PMID 20421958
- [Background] Murphy A, Kist C, Gier AJ, Edwards NM, Gao Z, Siegel RM. The feasibility of high-intensity interval exercise in obese adolescents. Clin Pediatr (Phila). 2015 Jan;54(1):87-90. doi: 10.1177/0009922814528038. Epub 2014 Mar 24. No abstract available. PMID 24662421
- [Background] Howe CA, Freedson PS, Feldman HA, Osganian SK. Energy expenditure and enjoyment of common children's games in a simulated free-play environment. J Pediatr. 2010 Dec;157(6):936-942.e1-2. doi: 10.1016/j.jpeds.2010.06.041. Epub 2010 Aug 13. PMID 20708746
- [Background] Fernandes RA, Zanesco A. Early sport practice is related to lower prevalence of cardiovascular and metabolic outcomes in adults independently of overweight and current physical activity. Medicina (Kaunas). 2015;51(6):336-42. doi: 10.1016/j.medici.2015.10.003. Epub 2015 Nov 17. PMID 26739675
- [Background] Bendiksen M, Williams CA, Hornstrup T, Clausen H, Kloppenborg J, Shumikhin D, Brito J, Horton J, Barene S, Jackman SR, Krustrup P. Heart rate response and fitness effects of various types of physical education for 8- to 9-year-old schoolchildren. Eur J Sport Sci. 2014;14(8):861-9. doi: 10.1080/17461391.2014.884168. Epub 2014 Feb 18. PMID 24533471
- [Background] Janssen I, Leblanc AG. Systematic review of the health benefits of physical activity and fitness in school-aged children and youth. Int J Behav Nutr Phys Act. 2010 May 11;7:40. doi: 10.1186/1479-5868-7-40. PMID 20459784
- [Background] McNarry MA, Lambrick D, Westrupp N, Faulkner J. The influence of a six-week, high-intensity games intervention on the pulmonary oxygen uptake kinetics in prepubertal obese and normal-weight children. Appl Physiol Nutr Metab. 2015 Oct;40(10):1012-8. doi: 10.1139/apnm-2015-0051. Epub 2015 Jun 12. PMID 26352388
- [Background] Metcalf B, Henley W, Wilkin T. Effectiveness of intervention on physical activity of children: systematic review and meta-analysis of controlled trials with objectively measured outcomes (EarlyBird 54). BMJ. 2012 Sep 27;345:e5888. doi: 10.1136/bmj.e5888. PMID 23044984
- See also: Description Website that was used for the recruitment, currently under development to included the results and publication of the study — http://top.ulusofona.pt